CLINICAL TRIAL: NCT05318430
Title: Subcutaneous Closed-Suction Drainage Affects Surgical Wounds Healing in Lower Gastrointestinal Open Surgery: a Randomized Controlled Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Director, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFH-SCD
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: All Diseases That Require Gastrointestinal Open Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): the closed-suction drainage device will be placed subcutaneously when closing the incision
  Interventions: Device: Subcutaneous closed-suction drainage device
- Control group (No Intervention): the closed-suction drainage device will not be placed subcutaneously when closing the incision

INTERVENTIONS:
Device: Subcutaneous closed-suction drainage device — This subcutaneous closed-suction drainage device was designed to be placed subcutaneously when surgeons have completed all intra-abdominal operations and are about to suture subcutaneous layer and skin
  Arms: Experimental group

SUMMARY:
This is a single-center, randomized controlled trial to evaluate whether subcutaneous closed-suction drainage would decrease the incidence of poor surgical site healing in lower gastrointestinal open surgery. The independent risk factors of the incidence of poor surgical wounds healing in lower gastrointestinal open surgery will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-85 years old, male or female
* all patients underwent lower gastrointestinal surgery: the digestive tract below Treitz ligament was called lower gastrointestinal tract, including jejunum, ileum, ileocecal part and colorectal
* open surgery (instead of laparoscopic) required
* willing participated in clinical verification and signed informed consent.

Exclusion Criteria:

* laparoscopic surgery
* upper gastrointestinal surgery (esophagus, stomach, duodenum and hepatobiliary pancreas)
* simple appendectomy / total appendectomy
* hernia surgery and intestinal obstruction surgery without intestinal resection
* infection of incision site before operation
* pregnant women
* expected death within 1 month after operation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of poor healing of incisions | Within 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Export of individual patient data is not permitted by Chinese laws